CLINICAL TRIAL: NCT02672917
Title: Phase 1 Safety and Tolerability Study of Human Monoclonal Antibody 5B1 (MVT-5873) With Expansion in Subjects With Pancreatic Cancer or Other CA19-9 Positive Malignancies
Brief Title: Study of HuMab-5B1 (MVT-5873) in Subjects With Pancreatic Cancer or Other Cancer Antigen 19-9 (CA19-9) Positive Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: BioNTech Research & Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: BioNTech SE (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MV-0715-CP-001.01
Record Dates: First submitted 2016-01-25; First posted 2016-02-03 (Estimated); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Pancreatic Cancer
Keywords: CA19-9 Positive Malignancies; Pancreatic Cancer and other CA19-9 expressing malignancies; Pancreatic Ductal Adenocarcinoma (PDAC); Sialyl Lewis A (sLea)
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (6):
- Group A (Experimental): MVT-5873 monotherapy dose escalation, initial to MTD
  Interventions: Drug: MVT-5873
- Group B (Experimental): MVT-5873 is administered in Group B every 1 week in combination with gemcitabine and nab-paclitaxel
  Interventions: Drug: MVT-5873; Drug: gemcitabine + nab-paclitaxel
- Group C (Experimental): MVT-5873 is administered in Group C every 4 weeks by intravenous infusion following a lead in dose. Each cycle is 28 days. During dose escalation, doses of MVT-5873 will be increased to define the MTD. Up to 30 patients will be treated at the RP2D.
  Interventions: Drug: MVT-5873
- Group D (Experimental): MVT-5873 is administered in Group D every 2 weeks by intravenous infusion following a lead in dose. During dose escalation, doses of MVT-5873 will be increased to defined the MTD. Up to 30 patients will be treated at the RP2D.
  Interventions: Drug: MVT-5873
- Group E - metastatic (Experimental): MVT-5873 is administered in combination with mFOLFIRINOX every 2 weeks. Both MVT-5873 and mFOLFIRINOX will be administered by intravenous infusion. During dose escalation, doses of MVT-5873, will be increased to define the MTD in combination with mFOLFIRINOX. mFOLFIRINOX will be administered according to institutional standards in compliance with the package insert for each drug. Up to 30 patients will be treated at the RP2D.
  Interventions: Drug: MVT-5873; Drug: modified FOLFIRINOX (mFOLFIRINOX)
- Group F - adjuvant (Experimental): MVT-5873 is administered in combination with mFOLFIRINOX every 2 weeks. Both MVT-5873 and mFOLFIRINOX will be administered by intravenous infusion. During dose escalation, doses of MVT-5873, will be increased to define the MTD in combination with mFOLFIRINOX. mFOLFIRINOX will be administered according to institutional standards in compliance with the package insert for each drug. Up to 30 patients will be treated at the RP2D.
  Interventions: Drug: MVT-5873; Drug: modified FOLFIRINOX (mFOLFIRINOX)

INTERVENTIONS:
Drug: MVT-5873 — intravenous infusion (IV)
  Other Names: HuMab-5B1
Drug: modified FOLFIRINOX (mFOLFIRINOX) — IV
  Arms: Group E - metastatic; Group F - adjuvant
Drug: gemcitabine + nab-paclitaxel — IV
  Arms: Group B

SUMMARY:
Phase 1 Safety and Tolerability Study in Subjects with Pancreatic Cancer or Other CA19-9 Positive Malignancies.

DETAILED DESCRIPTION:
Open label, multicenter, non-randomized, dose escalation/expansion trial of MVT-5873 as a single agent and in combination with standard of care chemotherapy or modified FOLFIRINOX (mFOLFIRINOX) in subjects with pancreatic and other CA19-9 positive malignancies. The study was designed to define a Maximum Tolerated Dose (MTD) of MVT-5873 as monotherapy (Group A), in combination with a standard of care chemotherapy (Group B), for a Q2 week schedule (Group D), an MTD of MVT-5873 for a Q4 week schedule (Group C), and an MTD for a Q2 week schedule of MVT-5873 in combination with mFOLFIRINOX (Groups E and F). Each group utilized a conventional 3+3 study design to identify the MTD and recommended phase 2 dose (RP2D).

Following the definition of the MTD in each group, the RP2D of MVT-5873 as a single agent and in combination with mFOLFIRINOX was defined. Following completion of monotherapy dose escalation, an expansion cohort of 30 additional subjects was treated at the RP2D for Group D. Subjects were subdivided into two groups of 15 subjects; those without peripheral blood expression of C19-9 and those with peripheral blood expression of CA19-9. MVT-5873 pharmacokinetics (PK) and pharmacodynamics (PD) were determined for each group.

ELIGIBILITY:
Inclusion Criteria [all groups]

* Signed, informed consent
* Age 18 or more years
* Histologically or cytologically confirmed, locally-advanced or metastatic pancreatic ductal adenocarcinoma (PDAC) or other CA19-9 positive malignancies
* Recovered from prior treatment related toxicity to at least Grade 1 with exception of Grade 2 alopecia or other Grade 2 toxicity with approval of the Medical Monitor
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1 or KPS of 100% to 80%
* Adequate hematologic, hepatic, and renal function
* Willingness to participate in collection of pharmacokinetic samples
* Willingness to use adequate contraception throughout study and for a period of 3 months after last dose of MVT-5873 and for up to at least 9 months after the last Oxaliplatin dose.

[Group A, C, and Group D Dose Escalation]

* Evaluable or measurable disease based on RECISTv1.1

[Group A, C, and D]

* Progression following treatment with standard of care for the subject's specific tumor type

[Group C and D Dose Expansion and Group E Dose Escalation and Expansion]

* Measurable disease based on RECISTv1.1

[Group C and D Dose Expansion, non-PDAC malignancies]

* If serum CA19-9 levels (defined as < 1 U/mL or below the level of detection for institutional test used), subject must have confirmation of CA19-9 expression in their tumor prior to study entry (based on institutional determination of CA19-9)

[Group E and F]

* Candidates for mFOLFIRINOX based on accepted standard of care

[Group F]

* Histologically or cytologically confirmed PDAC
* Macroscopically complete resection (R0 or R1 resection) performed between ≥21 and ≤84 days prior to Cycle 1, Day 1 (C1D1)
* Baseline scans without evidence of disease (e.g., CT/MRI)
* Serum CA19-9 ≤ 180 U/mL within 21 days of C1D1
* Full recovery from surgery and able to receive chemotherapy
* Free of significant nausea and vomiting
* No prior radiotherapy or chemotherapy

Exclusion Criteria [Groups A, B, C, D, and E]

* Brain metastases unless previously treated and well controlled for at least 3 months prior to study day 1
* Other known active cancer(s) likely to require treatment in the next two (2) years
* Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy
* Fewer than 28 days (or 5 half-lives for systemic agents, whichever is shorter) from prior anticancer therapy including chemotherapy, hormonal, investigational, and/or biological therapies and irradiation (except for ongoing hormonal therapy for prostate cancer)
* Major surgery within 28 days of Study Day 1
* History of anaphylactic reaction to human, or humanized, antibody
* Pregnant or currently breast-feeding
* Known HIV, Hepatitis B or C-positive
* Psychiatric illness/social situations that would interfere with compliance with study requirements
* Significant cardiovascular risk (e.g., coronary stenting within 4 weeks, myocardial infarction within 6 months)

[Group F]

* Incomplete macroscopic tumor removal (R2 resection)
* Other known active cancer(s) likely to require treatment in the next 2 years
* Active, uncontrolled bacterial, viral, or fungal infection (s) requiring systemic therapy
* History of anaphylactic reaction to human, or humanized, antibody
* Pregnant or currently breast-feeding
* Known HIV, Hepatitis B or C-positive
* Psychiatric illness/social situations that would interfere with compliance with study requirements
* Significant cardiovascular risk (e.g., coronary stenting within 4 weeks, myocardial infarction within 6 months)
* Pre-existing neuropathy
* Known homozygous for UGT1A1*28 mutation
* Inflammatory disease of the colon or rectum, or occlusion or sub-occlusion of the intestine or severe postoperative uncontrolled diarrhea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
Group D - Determine the safety (treatment related adverse events as assessed by Common Toxicity Criteria for Adverse Events [CTCAE] V5.0) of MVT-5873 on a Q2 week schedule | Through study completion. Estimated at one year
Group D - Determine the MTD and/or RP2D of MVT-5873 on a Q2 week schedule | Through study completion. Estimated at one year
Group E - Determine the safety (treatment related adverse events as assessed by CTCAE V5.0) of MVT-5873 in combination with the modified FOLFIRINOX regimen (mFOLFIRINOX) in the metastatic disease setting | Through study completion. Estimated at one year
Group E - Determine the MTD and/or the RP2D of MVT-5873 in combination with the modified FOLFIRINOX regimen (mFOLFIRINOX) in the metastatic disease setting | Through study completion. Estimated at one year
Group F - Determine the safety (treatment related adverse events as assessed by CTCAE V5.0) of MVT-5873 in combination with the modified FOLFIRINOX regimen (mFOLFIRINOX) in the PDAC adjuvant setting | Through study completion. Estimated at one year
Group F - Determine the MTD and/or the RP2D of MVT-5873 administered in combination with the modified FOLFIRINOX regimen (mFOLFIRINOX) in the PDAC adjuvant setting | Through study completion. Estimated at one year

SECONDARY OUTCOMES:
Group D - Evaluate the hepatic safety profile (treatment related adverse events as assessed by CTCAE V5.0) of MVT-5873 in participants without elevated circulating CA19-9 expression | Through study completion. Estimated at one year
All groups - Evaluate pharmacokinetics (PK): Area Under the Curve (AUC) for MVT-5873 | Through study completion. Estimated at one year
  Determined using non-compartmental model.
All groups - Evaluate PK: Maximum concentration (Cmax) for MVT-5873 | Through study completion. Estimated at one year
  Determined using non-compartmental model.
All groups - Evaluate PK: Plasma half-life (T1/2) for MVT-5873 | Through study completion. Estimated at one year
  Determined using non-compartmental model.
Groups A, B, C, D, E - Evaluate tumor response rate | Through study completion. Estimated at one year
Groups A, B, C, D, E - Evaluate duration of response | Through study completion. Estimated at one year
Groups A, B, C, D, E - Evaluate time to response | Through study completion. Estimated at one year
Groups A, B, C, D, E - Evaluate progression free survival | Through study completion. Estimated at one year
All groups - Evaluate overall survival | Through study completion. Estimated at one year
Group F - Evaluate disease free survival | Through study completion. Estimated at one year
Group F - Evaluate time to recurrence | Through study completion. Estimated at one year

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (5):
- United States (5):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - The Angeles Clinic & Research Institute, Los Angeles, California
  - Florida Cancer Specialist and Research Institute, Sarasota, Florida
  - MSKCC, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No